CLINICAL TRIAL: NCT02110147
Title: Open-Label Study of Uridine Triacetate in Pediatric Patients With Hereditary Orotic Aciduria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wellstat Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 401.13.001
Record Dates: First submitted 2014-04-01; First posted 2014-04-10 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-06

CONDITIONS: Hereditary Orotic Aciduria
MeSH Terms: conditions — Oroticaciduria 1 | interventions — uridine triacetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Uridine Triacetate to Replace Uridine (Experimental): Replacement therapy for oral uridine with oral administration of uridine triacetate in patients with hereditary orotic aciduria who have received (or would reasonably be expected to receive) clinical benefit from treatment with exogenous uridine. The starting dose of uridine triacetate will be 60 mg/kg/day which may be escalated to 300 mg/kg/day of oral uridine triacetate. The dose may be given once a day or as equally divided doses twice a day.
  Interventions: Drug: uridine triacetate

INTERVENTIONS:
Drug: uridine triacetate
  Other Names: PN401 (Company Code Name); 2',3',5'-tri-O-acetyluridine

SUMMARY:
This protocol has two parts - the Main Study which is 42 days in length and the Treatment Extension which allows the patients who complete the Main Study to continue receiving treatment with uridine triacetate. The purpose of this study is to replace oral administration of uridine with oral administration of uridine triacetate in patients with hereditary orotic aciduria who have received (or would reasonably be expected to receive) clinical benefit from treatment with exogenous uridine. It is also to document the continued clinical benefit of exogenous uridine when patients are switched from oral administration of uridine to oral administration of uridine triacetate.

DETAILED DESCRIPTION:
Data to be collected during the Main Study include demographic, baseline disease information and medical history including all prior disease-directed therapy. In addition, vital signs, laboratory values and adverse events information will be collected and recorded. Urine samples will be obtained and measured for orotic acid and orotidine levels. Systemic levels of uridine will be evaluated from plasma samples collected at set timepoints.

Upon successful completion of the Main Study and entry into the Treatment Extension, physical exams and vital signs will be performed every six (6) months. Additionally, plasma samples to measure systemic levels of uridine and urine samples to measure levels of orotic acid and orotidine will be collected every (6) six months.

ELIGIBILITY:
Inclusion Criteria (Main Study):

* Patients with diagnosed hereditary orotic aciduria
* Judged by the investigator to have the initiative and means to be compliant with the protocol
* Able to take oral medications
* Able to provide written informed consent (patient or legally authorized representative)
* Females of childbearing potential must have a negative pregnancy test at screening
* Females of childbearing potential or males with partners of childbearing potential are to use one of the following acceptable birth control methods:
* Surgically sterile or partner is surgically sterile
* Using adequate contraception (hormonal contraceptives, double barrier methods, or intra-uterine devices)
* Patients who claim to be sexually inactive agree to use an acceptable method of contraception should she or he become sexually active from 14 days prior to first dosing, throughout the study and for 14 days after the last dose administration

Exclusion Criteria (Main Study):

* Has a known allergy to uridine triacetate or any of its excipients
* Known to have ornithine transcarbamoylase deficiency
* Unable to have the initiative and means to be compliant with the protocol
* Unable to be compliant with taking oral medications
* Unable to provide written informed consent (patient or legally authorized representative)
* Female who is pregnant or lactating

Inclusion Criteria (Treatment Extension)

* Patient successfully completed the Main Study

Exclusion Criteria (Treatment Extension)

* Patient did not successfully complete the Main Study

Ages: 6 Months to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2016-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael K. Bamat, Ph.D., Study Director — Wellstat Therapeutics
Locations (2):
- United States (2):
  - Children's Hospital of Michigan - Specialty Center Detroit, Detroit, Michigan
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: All patients were treated with uridine triacetate oral granules.
Period: Overall Study
Arm/Group | Single Arm
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Patients With Stable Predetermined Principal Hematologic Parameters
Description: Hereditary orotic aciduria patients will be taking uridine triacetate as replacement therapy for uridine. The primary outcome measure will be based on predetermined principal hematologic parameter(s) based on the patient's response(s) to oral uridine when dosing is switched from oral uridine to oral uridine triacetate. The primary outcome measure in patients not previously receiving uridine replacement therapy will be improvement in the patient's principal affected hematologic parameter(s) on Days 28 and 42 compared to baseline (Day 0) of the Main Study.
Time Frame: Days 28 and 42
Measure: Count of Participants; unit: Participants
Groups:
- Uridine Triacetate: All patients were treated with uridine triacetate oral granules.
Arm/Group | Uridine Triacetate
Number analyzed (Participants) | 4
Participants | 4

2. Secondary Outcome: Patients With Stable or Improved Orotic Acid and Orotidine Levels
Description: Significantly elevated urine orotic acid levels are characteristic of patients with HOA. Therefore, urinary orotic acid and orotidine levels were assessed in patients at baseline (on uridine or uridine naïve) and on Day 28 and Day 42 following the switch to uridine triacetate. The table below shows the number of participants with stable or improved orotic acid and orotidine levels at Day 28 and Day 42 compared to baseline.
Time Frame: Days 28 and 42
Measure: Count of Participants; unit: Participants
Arm/Group | Uridine Triacetate
Number analyzed (Participants) | 4
Participants
  Day 28 | 4
  Day 42 | 4

3. Secondary Outcome: Patients With Levels of Uridine in the Plasma Consistent With Expected Therapeutic Benefit
Description: HOA is principally a chronic uridine deficiency disorder. The purpose of uridine triacetate administration is to provide an exogenous source of uridine. Therefore, plasma uridine levels were assessed at various time points (prior to dosing, 30 min, 1 hour, 2 hours, 4 hours, 6 hours and 8 hours) following uridine triacetate dosing to ensure levels of uridine consistent with previously observed symptomatic improvement from administration of uridine were achieved. The table below shows the number of participants with uridine levels consistent with or exceeding previously observed symptomatic improvements.
Time Frame: Days 1 and 28
Measure: Count of Participants; unit: Participants
Arm/Group | Uridine Triacetate
Number analyzed (Participants) | 4
Participants
  Day 1 | 4
  Day 28 | 4

ADVERSE EVENTS:
Time Frame: Safety data collected for 24 months.
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No